CLINICAL TRIAL: NCT04043377
Title: 68Ga-DOTATATE PET-CTA Imaging for the Early Detection of Progressing Coronary Atherosclerosis
Acronym: iPROGRESS
Status: Terminated | Phase: Phase 3 | Type: Interventional
Why Stopped: Financial issues
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: P 171103; 2017-004793-34 (EudraCT Number)
Record Dates: First submitted 2019-07-23; First posted 2019-08-02 (Actual); Last update posted 2022-06-30 (Actual); Status verified 2022-06

CONDITIONS: Coronary Arteriosclerosis
Keywords: Coronary atherosclerosis; 68Ga-DOTATATE; PET-CTA imaging; No significant myocardial ischemia
MeSH Terms: conditions — Coronary Artery Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- All patients (Experimental)
  Interventions: Drug: injection of 68Ga-DOTATATE

INTERVENTIONS:
Drug: injection of 68Ga-DOTATATE — PET after injection of 68Ga-DOTATATE 2 MBq/kg (Max. 200 MBq); intra-venous; single injection, at M0 followed by a coronary CTA to localize the signal in coronary arteries Consultation and low-dose cardiac CT for coronary calcium scoring performed at M12 and M24 after inclusion.

SUMMARY:
68Ga-DOTATATE is a PET radiotracer with high affinity and selectivity for somatostatin receptor 2 (SSTR 2) and is approved clinically for the evaluation of patients with neuroendocrine tumors. The SSTR2 receptor is also highly expressed at the surface of human macrophages and lymphocytes. In comparison to FDG, 68Ga-DOTATATE presents the advantage of fast clearance from tissues, which are not expressing somatostatin receptors, in particular muscular and myocardial tissues, and the level of blood glucose does not influence its uptake.

Accumulation of 68Ga-DOTATATE has already been detected in coronary and carotid plaques and is associated with the number of activated macrophages present in plaques obtained after carotid endarterectomy. In a recent study, Tarkin et al. confirmed the preferential uptake of 68Ga-DOTATATE by macrophages in atherosclerotic plaques. In addition, the intensity of 68Ga-DOTATATE was higher in culprit lesions in the carotid and coronary arteries than in stable lesions. The evaluation of 68Ga-DOTATATE uptake in coronary arteries was also strongly facilitated in comparison to FDG thanks to the absence of spillover signal from the myocardium.

AAA has developed a new kit that has markedly simplified the synthesis of 68Ga-DOTATATE and has obtained in the US marketing authorization for the kit (Netspot; kit for the preparation of Gallium-68-DOTATATE injection for intravenous use) on June 1st 2016 (NDA 208547) for evaluation of patients with neuro-endocrine tumors. The Netspot kit will be used in this study for the detection of progressing coronary atherosclerosis.

DETAILED DESCRIPTION:
Design of the trial :

iPROGRESS is a prospective interventional study. The primary objective of this study will be to test the association between the intensity of 68Ga-DOTATATE uptake in coronary plaques quantified with PET at M0 and the absolute progression rate of coronary artery calcium scoring (CACS) measured between the CT acquired at M0 and after 2 years.

Patients will be screened until 1 month before the inclusion (M0) visit. Thereafter, 3 visits specifics to the study will be performed.

M0 (baseline): Injection of 68Ga-DOTATATE followed by PET-scan and a CCTA-scan M12 et M24(follow-up): Consultation and low-dose cardiac CT for coronary calcium scoring performed

ELIGIBILITY:
Inclusion Criteria:

* Patients with a coronary artery calcium score (CACS) measured with a low-dose CT between 100 and 1000 and absence of significant ischemia (≥ 12 % of the myocardium) on myocardial perfusion scintigraphy.
* Age ≥ 18 years
* Affiliation to a social security regime
* Signed informed consent.

Exclusion Criteria:

Exclusion Criteria :

* Previous acute coronary syndrome or coronary revascularisation
* LVEF < 40 %
* Previous severe adverse reaction to iodinated contrast agent
* Irregular heart rhythm (chronic atrial fibrillation, numerous extrasystoles)
* Severe asthma
* Chronic kidney disease (eGFR < 45 ml/min/1.73 m2)
* Waldenstrom disease
* Multiple myeloma
* Autoimmune / inflammatory disease requiring immunosuppressive treatment.
* Active cancer.
* Confirmed or suspected pregnancy
* Breast feeding
* Impossibility to stay immobile and maintain the supine position during 30 minutes.
* Patient deprived of liberty or under legal protection measure
* Participation to an interventional trial involving the use of radiation during the two years of the study.
* Participation to an interventional trial with the use of new drugs between the inclusion and one month after injecting 68Ga-DOTATATE.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2019-11-21 (Actual); Primary Completion 2021-09-13 (Actual); Study Completion 2021-09-13 (Actual)

PRIMARY OUTCOMES:
Absolute increase in calcium artery calcium scoring (CACS) per year. | 2 years
  The volume of calcium along coronary arteries will be measured on low-dose gated CT acquisitions using a dedicated software. The increase in CACS will be measured as the difference between the CACS measured at baseline and 2 years later and a yearly increase rate of CACS will be calculated.

SECONDARY OUTCOMES:
Combined end point including cardiovascular death, acute coronary syndrome and ischemia-driven coronary revascularization. | 2 years
  Two years after the inclusion, the patient will be interviewed for the occurrence of cardiovascular events. In case of a suspicion of cardiovascular event, the report of the hospital will be collected or the physician in charge of the patient will be contacted.
Characterization of coronary plaques 1 | 2 years
  Coronary CTA will be analysed using a dedicated software. Each coronary plaque detected on the CCTA will be characterized as:
  * non-calcified
  * mixed
  * calcified High-risk plaques will be defined on CCTA as non-calcified plaque with hypodense region and positive remodelling.
Characterization of coronary plaques 2 | 2 years
  Coronary CTA will be analysed using a dedicated software. Each coronary plaque detected on the CCTA will be characterized as:
  * presence of hypodense region
  * absence of hypodense region (< 30 HU), High-risk plaques will be defined on CCTA as non-calcified plaque with hypodense region and positive remodelling.
Characterization of coronary plaques 3 | 2 years
  Coronary CTA will be analysed using a dedicated software. Each coronary plaque detected on the CCTA will be characterized by: maximal plaque surface.
  High-risk plaques will be defined on CCTA as non-calcified plaque with hypodense region and positive remodelling.
Characterization of coronary plaques 4 | 2 years
  Coronary CTA will be analysed using a dedicated software. Each coronary plaque detected on the CCTA will be characterized by: plaque remodelling ratio.
  High-risk plaques will be defined on CCTA as non-calcified plaque with hypodense region and positive remodelling.
Characterization of coronary plaques 5 | 2 years
  Coronary CTA will be analysed using a dedicated software. Each coronary plaque detected on the CCTA will be characterized by: degree of luminal stenosis (%).
  High-risk plaques will be defined on CCTA as non-calcified plaque with hypodense region and positive remodelling.
MDS TBR of coronary arteries and global TBR of the thoracic aorta. | 2 years
  The most-diseased segment (MDS) will be defined as the max. TBR value with the highest signal along coronary arteries for each patient. Global TBR of the thoracic aorta will be calculated as the average of max. TBR measured on 2D ROI placed on the thoracic aorta.
68Ga-DOTATATE uptake in the parodontal bone. | 2 years
  The intensity of 68Ga-DOTATATE uptake in periodontal bone will be measured on the PET acquired at M0 as average of four TBR max. values measured in each quadrant of the mouth.

CONTACTS AND LOCATIONS:
Overall Officials: Fabien HYAFIL, Doctor, Principal Investigator — Assistance Publique - Hôpitaux de Paris
Locations (1):
- service de médecine nucléaire-Hôpital Bichat, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided